CLINICAL TRIAL: NCT03981653
Title: Angiogenic Function at Normal Term on Placenta
Acronym: ANNOTEP
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANNOTEP
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In vivo and ex vivo study of trophoblastic angiogenic trophoblastic function in placentas from normal pregnancies, at term

DETAILED DESCRIPTION:
The objective of this study is to better understand the regulation of trophoblast expression of pro- and antiangiogenic factors such as placenta growth factor (PlGF) or Soluble FMS like tyrosin-kinase-1 (sFlt-1), and more particularly on human differentiated trophoblastic cells from "healthy" placentas. The measurement of the variation in gene and protein expression of placental angiogenic factors will provide a better understanding of their pathophysiology.

Secondary objectives are the study of trophoblastic differentiation and placental functions, and the study of the impact of chemical compounds on the biological functions of the placenta. To do this, these "healthy" placentas may be exposed to different factors that promote the occurrence of specific pregnancy pathologies such as pre-eclampsia and vascular intrauterine growth restriction (IUGR), caused by placental dysfunction. This will make it possible to test molecules and vector approaches targeted directly at the trophoblast, in order to consider therapeutic targets, which do not exist to date.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies with scheduled cesarean delivery >37 weeks of amenorrhea:
* strictly normal pregnancies
* complicated pregnancies of gestational diabetes, insulin-treated or not
* complicated pregnancies due to pregnancy cholestasis
* spontaneous or in vitro fecondation (IVF) / Intracytoplasmic sperm injection (ICSI) pregnancies with or without oocyte donation

Exclusion Criteria:

* Patient's opposition
* Age < 18 years old
* Women under the protection of justice
* Multiple pregnancy
* Known major fetal malformation
* Pre-eclampsia and intrauterine growth retardation
* Placental insertionnomaly
* Type 1 diabetes
* HIV-positive patient with HIV/hepatisis C virus (HCV) regardless of viral load
* Patient in labour at the time of Caesarean section
* Patient whose medical history results in medication being taken in pregnancy courses that may interfere with the biology of the trophoblast (immunomodulators in case of autoimmune diseases, anti-rejection drugs in case of transplant patients)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with a progressive, full-term pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Level of placental angiogenic factors | day 0
  Variation in the gene and protein expression of placental angiogenic factors on healthy placentas

SECONDARY OUTCOMES:
Level of sFlt-1 (Soluble FMS like tyrosin-kinase-1) | day 1
  Sflt-1 levels when the placenta is exposed to factors that promote the development of vascular pregnancy diseases
Level of PlGF (Placental Growth Factor) | day 1
  PlGF levels when the placenta is exposed to factors that promote the development of vascular pregnancy diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No